CLINICAL TRIAL: NCT04946877
Title: Clinical Study of Comorbidities of Attention Deficit Hyperactivity in Children and Adolescents.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Mohmed, Doctor, Assiut University
Other Study IDs: Comorbidities with ADHD
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD,comorbidities
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: 100 ADHD patients; will be taken from outpatient clinic of child and adolescence psychiatry of Assiut university hospitals.
  Interventions: Diagnostic Test: IQ assessment using Wechsler intelligence scale for children third edition (WISC-III)
- control group: 100 normal children; they will be selected from neurology clinic complaining from minor neurological complaint e.g : headache, will match with the case group for age, sex and educational level.
  Interventions: Diagnostic Test: IQ assessment using Wechsler intelligence scale for children third edition (WISC-III)

INTERVENTIONS:
Diagnostic Test: IQ assessment using Wechsler intelligence scale for children third edition (WISC-III) — IQ assessment using Wechsler intelligence scale for children third edition (WISC-III): is consists of several subtests, each classified into a verbal or performance scale .
  Other Names: Mini international neuropsychiatric interview for children and adolescents (M.I.N.I. Kid); Child behavior checklist (CBCL), parent form; Neurological assessment using Cambridge neurological inventory

SUMMARY:
Determine the frequency of psychiatric and neurological comorbidities in children and adolescence diagnosed with ADHD.

DETAILED DESCRIPTION:
ADHD is a common neurodevelopmental disorder characterized by hyperactivity, impulsivity, and inattention .ADHD is more often a complex disorder with a high rate of associated co-morbid conditions. Co-morbid conditions are prevalent among people with ADHD and increase its burden and complexity of management.Children with ADHD are at a higher risk than children without ADHD for developing other psychiatric disorders .Motor skill problems and Neurological soft signs are found in many neuropsychiatric conditions .NSS have been associated with inattention and behaviour difficulties for decades. Some researchers argue that these signs should be included in the diagnosis of ADHD .

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-17 years.
* Sex: both sexes will be included in the study.
* IQ≥70.

Exclusion Criteria:

* Age: less than 6 years or more than 17 years.
* IQ<70.
* Patients with major neurological deficits, cerebral palsy and uncontrolled epilepsy.
* Patients with major psychiatric disorders e.g schizophrenia spectrum disorder.
* Patient who refusing to participate in the study or their caregiver refusing to give informed consent.

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Case group will include 100 ADHD patients; will be taken from outpatient clinic of child and adolescence psychiatry of Assiut university hospitals.
  Control group will include 100 normal children; they will be selected from neurology clinic complaining from minor neurological complaint e.g : headache, will match with the case group for age, sex and educational level.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Determine psychiatric comorbidities in children and adolescents with ADHD using Mini international neuropsychiatric interview for children and adolescents (M.I.N.I. Kid). | baseline
  Mini international neuropsychiatric interview for children and adolescents (M.I.N.I. Kid): is structured clinical diagnostic interview designed to assess the presence of current ICD-10 and DSM-IV psychiatric disorders in children and adolescents age 6-17 years

SECONDARY OUTCOMES:
determinate presence of soft neurological sign in children and adolescents with ADHD using Cambridge neurological inventory. | baseline
  Neurological assessment using Cambridge neurological inventory: this is a clinical instrument constructed for standardized neurological assessment of psychiatric patients. It is useful for identifying neurological soft sign and other patterns of neurological impairments

REFERENCES:
- [Background] Gillberg C, Gillberg IC, Rasmussen P, Kadesjo B, Soderstrom H, Rastam M, Johnson M, Rothenberger A, Niklasson L. Co-existing disorders in ADHD -- implications for diagnosis and intervention. Eur Child Adolesc Psychiatry. 2004;13 Suppl 1:I80-92. doi: 10.1007/s00787-004-1008-4. PMID 15322959
- [Background] Faraone SV, Asherson P, Banaschewski T, Biederman J, Buitelaar JK, Ramos-Quiroga JA, Rohde LA, Sonuga-Barke EJ, Tannock R, Franke B. Attention-deficit/hyperactivity disorder. Nat Rev Dis Primers. 2015 Aug 6;1:15020. doi: 10.1038/nrdp.2015.20. PMID 27189265
- [Background] Jensen CM, Steinhausen HC. Comorbid mental disorders in children and adolescents with attention-deficit/hyperactivity disorder in a large nationwide study. Atten Defic Hyperact Disord. 2015 Mar;7(1):27-38. doi: 10.1007/s12402-014-0142-1. Epub 2014 Jun 19. PMID 24942707